CLINICAL TRIAL: NCT01373346
Title: Long Limb Roux-en Y Reconstruction After Gastrectomy As A Potential Cure for Type 2 Diabetes Mellitus in Non-Obese Gastric Cancer Patients - a Pilot Project to Validate a Prospective Randomized Control Trial
Brief Title: Safety and Efficacy of Long Limb Roux-en Y Reconstruction
Acronym: LoLiRoRe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Seung Ho Choi, Chief of surgery, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: seungho-1
Record Dates: First submitted 2011-06-13; First posted 2011-06-14 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Diabetes Mellitus Type 2 in Nonobese; Gastric Cancer
Keywords: type II diabetes; Gastric cancer; Long limb Roux-en Y
MeSH Terms: conditions — Stomach Neoplasms; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Long limb Roux-en Y reconstruction (Experimental): Long limb Roux-en Y reconstruction means that the length of Roux limb and biliopancreatic limb are longer than conventional reconstruction method after gastrectomy.
  Interventions: Procedure: Long limb Roux-en Y reconstruction

INTERVENTIONS:
Procedure: Long limb Roux-en Y reconstruction — After radical gastrectomy, the gastrointestinal tract was reconstructed by Roux-en-Y gastrojejunostomy or esophagojejunostomy. The jejunum was divided at approximately 100-120 cm distal to the ligament of Treitz and the distal limb of the jejunum was then anastomosed along the proximal gastric greater curvature or esophagus. The jejuno-jejunostomy was performed approximately 100 to 120 cm distal from the gastrojejunal or esophagojejunal anastomosis
  Other Names: modified Roux-en Y

SUMMARY:
We grafted the concept of metabolic surgery (long limb Roux-en Y reconstruction) into gastric cancer surgery. This study aimed to investigate the safety and efficacy of long limb Roux-en Y reconstruction after gastrectomy in non-obese type II diabetes with gastric cancer.

DETAILED DESCRIPTION:
Type II diabetes in the world is increasing rapidly, and it is known that patients with type II diabetes with morbid obesity that underwent bariatric surgery have resolution of impaired glucose metabolism.

In Asia, most type II diabetes are not morbidly obese and still, it is controversy whether metabolic surgery is effective or not in non-morbid obese patients. As life expectancy is increased, the number of patients with gastric cancer and T2DM is increased as well.

Recently, we studied the outcome of T2DM after gastrectomy and conventional reconstruction in non-obese gastric cancer patients.(Kim JW et al, World J Gastroenterol 2012;18:49) The study was a large-series retrospective study including about 400 patients and the result regarding DM improvement was not satisfactory. Based on our previous results, it is needed to find more effective way to resolve the type II diabetes in gastrectomized patients with gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed gastric cancer with potentially curable state
* Non-obese (Body mass index: less than 30 kg/m2)
* Have a history of Type 2 DM over 6 months (diagnosed by ADA criteria)

  1. HBA1c: more than 6.5 %, or Fasting glucose: more than 126 mg/dl (7.0mmol/L) or 2-h plasma glucose: more than 200mg/dl during an OGTT or classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose: more than 200mg/dl
  2. Anti-GAD antibody (-), Anti-islet antibody (-)
* C-peptide level: above 1ng/ml

Exclusion Criteria:

* Patient who receive non-curative operation
* Patient who have less than one year life expectancy
* Pregnant patient
* Acute inflammation status patient
* Chronic renal disease patient (Serum creatin level: more than 1.5mg/dl)
* Chronic liver disease patient (Serum AST or ALT level: more than twice of upper limit of normal range)
* Have a history of receiving medications such as dipeptidyl peptidase IV(DPP- IV) inhibitor or glucagon like peptide-I (GLP-I) analogue

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seung Ho Choi, M.D., Ph.D., Principal Investigator — Department of Surgery, Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul, Korea
Locations (1):
- GangNam Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Buchwald H, Estok R, Fahrbach K, Banel D, Jensen MD, Pories WJ, Bantle JP, Sledge I. Weight and type 2 diabetes after bariatric surgery: systematic review and meta-analysis. Am J Med. 2009 Mar;122(3):248-256.e5. doi: 10.1016/j.amjmed.2008.09.041. PMID 19272486
- [Background] Pories WJ, Swanson MS, MacDonald KG, Long SB, Morris PG, Brown BM, Barakat HA, deRamon RA, Israel G, Dolezal JM, et al. Who would have thought it? An operation proves to be the most effective therapy for adult-onset diabetes mellitus. Ann Surg. 1995 Sep;222(3):339-50; discussion 350-2. doi: 10.1097/00000658-199509000-00011. PMID 7677463
- [Background] Yoon KH, Lee JH, Kim JW, Cho JH, Choi YH, Ko SH, Zimmet P, Son HY. Epidemic obesity and type 2 diabetes in Asia. Lancet. 2006 Nov 11;368(9548):1681-8. doi: 10.1016/S0140-6736(06)69703-1. PMID 17098087
- [Background] FRIEDMAN MN, SANCETTA AJ, MAGOVERN GJ. The amelioration of diabetes mellitus following subtotal gastrectomy. Surg Gynecol Obstet. 1955 Feb;100(2):201-4. No abstract available. PMID 13238177
- [Background] ANGERVALL L, DOTEVALL G, TILLANDER H. Amelioration of diabetes mellitus following gastric resection. Acta Med Scand. 1961 Jun;169:743-8. doi: 10.1111/j.0954-6820.1961.tb07885.x. No abstract available. PMID 13683582
- [Background] Yang J, Li C, Liu H, Gu H, Chen P, Liu B. Effects of subtotal gastrectomy and Roux-en-Y gastrojejunostomy on the clinical outcome of type 2 diabetes mellitus. J Surg Res. 2010 Nov;164(1):e67-71. doi: 10.1016/j.jss.2010.07.004. Epub 2010 Jul 30. PMID 20863527
- [Background] Kim JW, Cheong JH, Hyung WJ, Choi SH, Noh SH. Outcome after gastrectomy in gastric cancer patients with type 2 diabetes. World J Gastroenterol. 2012 Jan 7;18(1):49-54. doi: 10.3748/wjg.v18.i1.49. PMID 22228970
- [Background] DeFronzo RA, Matsuda M. Reduced time points to calculate the composite index. Diabetes Care. 2010 Jul;33(7):e93. doi: 10.2337/dc10-0646. No abstract available. PMID 20587713
- [Background] Emoto M, Nishizawa Y, Maekawa K, Hiura Y, Kanda H, Kawagishi T, Shoji T, Okuno Y, Morii H. Homeostasis model assessment as a clinical index of insulin resistance in type 2 diabetic patients treated with sulfonylureas. Diabetes Care. 1999 May;22(5):818-22. doi: 10.2337/diacare.22.5.818. PMID 10332688
- [Background] Katz A, Nambi SS, Mather K, Baron AD, Follmann DA, Sullivan G, Quon MJ. Quantitative insulin sensitivity check index: a simple, accurate method for assessing insulin sensitivity in humans. J Clin Endocrinol Metab. 2000 Jul;85(7):2402-10. doi: 10.1210/jcem.85.7.6661. PMID 10902785
- [Background] Frenken M, Cho EY, Karcz WK, Grueneberger J, Kuesters S. Improvement of type 2 diabetes mellitus in obese and non-obese patients after the duodenal switch operation. J Obes. 2011;2011:860169. doi: 10.1155/2011/860169. Epub 2011 Mar 3. PMID 21461399
- [Background] Navarrete SA, Leyba JL, Llopis SN. Laparoscopic sleeve gastrectomy with duodenojejunal bypass for the treatment of type 2 diabetes in non-obese patients: technique and preliminary results. Obes Surg. 2011 May;21(5):663-7. doi: 10.1007/s11695-011-0371-8. PMID 21336559
- [Background] Cohen R, Pinheiro JS, Correa JL, Schiavon CA. Laparoscopic Roux-en-Y gastric bypass for BMI < 35 kg/m(2): a tailored approach. Surg Obes Relat Dis. 2006 May-Jun;2(3):401-4, discussion 404. doi: 10.1016/j.soard.2006.02.011. PMID 16925363
- [Background] DePaula AL, Macedo AL, Mota BR, Schraibman V. Laparoscopic ileal interposition associated to a diverted sleeve gastrectomy is an effective operation for the treatment of type 2 diabetes mellitus patients with BMI 21-29. Surg Endosc. 2009 Jun;23(6):1313-20. doi: 10.1007/s00464-008-0156-x. Epub 2008 Oct 2. PMID 18830750
- [Background] Cohen RV, Schiavon CA, Pinheiro JS, Correa JL, Rubino F. Duodenal-jejunal bypass for the treatment of type 2 diabetes in patients with body mass index of 22-34 kg/m2: a report of 2 cases. Surg Obes Relat Dis. 2007 Mar-Apr;3(2):195-7. doi: 10.1016/j.soard.2007.01.009. No abstract available. PMID 17386401
- [Background] Orci L, Chilcott M, Huber O. Short versus long Roux-limb length in Roux-en-Y gastric bypass surgery for the treatment of morbid and super obesity: a systematic review of the literature. Obes Surg. 2011 Jun;21(6):797-804. doi: 10.1007/s11695-011-0409-y. PMID 21479976
- [Background] Rubino F, Forgione A, Cummings DE, Vix M, Gnuli D, Mingrone G, Castagneto M, Marescaux J. The mechanism of diabetes control after gastrointestinal bypass surgery reveals a role of the proximal small intestine in the pathophysiology of type 2 diabetes. Ann Surg. 2006 Nov;244(5):741-9. doi: 10.1097/01.sla.0000224726.61448.1b. PMID 17060767
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542

RESULTS

PARTICIPANT FLOW:
Recruitment Details: If Patients were eligible for the study, each patient was informed of the investigational nature of the trial and received detailed information regarding the study protocol. All patients provided written informed consent before their enrollment. The enrollment continued from February 2010 through May 2011 in Gangnam Severance Hospital.
Groups:
- Long Limb Roux-en Y Reconstruction: Total or Subtotal gastrectomized gastric cancer patient with long limb Roux en Y reconstruction
Period: Overall Study
Arm/Group | Long Limb Roux-en Y Reconstruction
Started | 15
Completed | 14
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Long Limb Roux-en Y Reconstruction
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 62.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 15

OUTCOME MEASURES:

1. Secondary Outcome: Matsuda Index
Description: Matsuda Index(Insulin Sensitivity Index) was measured.
  The Matsuda index was obtained using the following formula:
  Matsuda index = 10000/square root of [(fasting glucose × fasting insulin) × (mean glucose × mean insulin during OGTT)]
Time Frame: Before operation , 6 months after operation, Until end of study (on average 14.8 months)
Population: Fifteen patients were enrolled for this study. During the follow-up period, there was one patient, who had poorly differentiated neuroendocrine carcinoma which is one of most aggressive gastric cancer, and died due to recurrence four months after surgery. The patient who died of recurrence was excluded from the efficacy evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Long Limb Roux-en Y Reconstruction: Long limb Roux-en Y reconstruction means that the length of Roux limb and biliopancreatic limb are longer than conventional reconstruction method after gastrectomy. Briefly, the gastrointestinal tract was reconstructed by Roux-en Y gastrojejunostomy or esophagojejunostomy after radical gastrectomy. The jejunum was divided at approximately 100-120 cm distal to the ligament of Treitz and the distal limb of the jejunum was then anastomosed along the proximal gastric greater curvature or esophagus. The jejuno-jejunostomy was performed approximately 100 to 120 cm distal from the gastrojejunal or esophagojejunal anastomosis.
Arm/Group | Long Limb Roux-en Y Reconstruction
Number analyzed (Participants) | 14
units on a scale
  Before operation | 7.2 (5.0)
  6 months after operation | 15.4 (10.9)
  Until end of study (on average 14.8 months) | 17.1 (10.5)

2. Primary Outcome: Morbidity
Description: For the evaluation of safety, morbidity were analyzed. For the evaluation of short-term safety, complications higher than the Clavien-Dindo grade II (Dindo et. Ann Surg 240:205 2004) were collected.
  *Clavien-dindo classification of surgical complications Grade II: Requiring pharmacological treatment with drugs other than such allowed for grade I complications. Blood transfusions and total parenteral nutrition are also included.
  Grade III: Requiring surgical, endoscopic or radiological intervention Grade IV:Life-threatening complication (including CNS complications)‡ requiring IC/ICU-management Grade V:Death of a patient Suffix'd' : If the patient suffers from a complication at the time of discharge ,the suffix "d" (for 'disability') is added to the respective grade of complication. This label indicates the need for a follow-up to fully evaluate the complication.
  For the evaluation of long-term safety, the patients were evaluated every month after discharge.
Time Frame: Until end of study (on average 14.8 months)
Population: All of enrolled patient were included. (N=15)
Measure: Number; unit: participants
Groups:
- Long Limb Roux-en Y Reconstruction: Morbidity after operation were analyzed until end of study (on average 14.8 months)
Arm/Group | Long Limb Roux-en Y Reconstruction
Number analyzed (Participants) | 15
participants | 4

3. Secondary Outcome: QUICKI
Description: The quantitative insulin sensitivity check index (QUICKI) was measured.
  The QUICKI was obtained using the following formula:
  1 / (log(fasting insulin µU/mL) + log(fasting glucose mg/dL))
Time Frame: Before operation , 6 months after operation , Until end of study (on average 14.8 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Long Limb Roux-en Y Reconstruction
Number analyzed (Participants) | 14
units on a scale
  Pre Operation | 0.4 (0.1)
  6 months after operation | 0.4 (0.0)
  Until end of study (on average 14.8 months) | 0.4 (0.1)

4. Secondary Outcome: HOMA-IR
Description: HOMA-IR(Homeostasis model assessment-estimated insulin resistance) was measured.
  HOMA-IR was obtained using the following formula:
  Glucose(mg/dl) x Insulin/405
Time Frame: Before operation , 6 months after operation, Until end of study (on average 14.8 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Long Limb Roux-en Y Reconstruction
Number analyzed (Participants) | 14
units on a scale
  Before operation | 2.2 (2.4)
  6 months after operation | 1.0 (0.8)
  Until End of study(on average 14.8 months) | 1.0 (0.8)

5. Secondary Outcome: HOMA-B
Description: HOMA-B(Homoeostasis model assessment-derived beta-cell function) was measured.
  HOMA-B was obtained using the following formula:
  225 × 18/fasting insulin(mU/L) × fasting glucose(mg/dL)
Time Frame: Before operation , 6 months after operation, Until end of study (on average 14.8 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of beta cell function
Groups:
- Long Limb Roux en Y Reconstruction: Long limb Roux-en Y reconstruction means that the length of Roux limb and biliopancreatic limb are longer than conventional reconstruction method after gastrectomy. Briefly, the gastrointestinal tract was reconstructed by Roux-en Y gastrojejunostomy or esophagojejunostomy after radical gastrectomy. The jejunum was divided at approximately 100-120 cm distal to the ligament of Treitz and the distal limb of the jejunum was then anastomosed along the proximal gastric greater curvature or esophagus. The jejuno-jejunostomy was performed approximately 100 to 120 cm distal from the gastrojejunal or esophagojejunal anastomosis.
Arm/Group | Long Limb Roux en Y Reconstruction
Number analyzed (Participants) | 14
percentage of beta cell function
  Before operation | 7.7 (7.1)
  6 months after operation | 13.4 (8.1)
  Until end of study (on average 14.8 months) | 16.0 (11.1)

6. Secondary Outcome: Body Mass Index
Description: BMI(Body Mass index , kg/㎡) was measured.
  BMI was obtained using the following formula:
  Weight (kg) / (Height (m) x Height (m))
Time Frame: Before operation, 6 Months After Operation, Until End of Study(on Average 14.8 Months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/㎡
Arm/Group | Long Limb Roux en Y Reconstruction
Number analyzed (Participants) | 14
kg/㎡
  Before operation | 25.2 (3.4)
  6 months after operation | 21.7 (3.1)
  Until end of study (on average 14.8 months) | 21.2 (2.8)

7. Primary Outcome: HbA1c
Description: For the evaluation of efficacy for the operation, HbA1c(%) was measured serially (preop. 6months after op. until end of study(on average 14.8 months)).
  HbA1c is formed in a non-enzymatic glycation pathway by hemoglobin's exposure to plasma glucose and measured by high-performance liquid chromatography (HPLC) The HbA1c was calculated as a ratio to total hemoglobin.
Time Frame: Before operation , 6 months after operation, Until end of study (on average 14.8 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Long Limb Roux en Y Reconstruction
Number analyzed (Participants) | 14
percentage of glycated hemoglobin
  Before operation | 7.7 (1.4)
  6 months after operation | 6.3 (0.8)
  Until end of study (on average 14.8 months) | 6.3 (0.8)

8. Primary Outcome: Hemoglobin
Description: For the evaluation of long-term safety, hemoglobin was measured to determine the degree of anemia and malnutrition.
Time Frame: Before operation , 6 months after operation, Until end of study (on average 14.8 months)
Population: Fifteen patients were enrolled for this study. During the follow-up period, there was one patient, who had poorly differentiated neuroendocrine carcinoma which is one of most aggressive gastric cancer, and died due to recurrence four months after surgery. The patient who died of recurrence was excluded from the long-term safety evaluation.
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Long Limb Roux en Y Reconstruction
Number analyzed (Participants) | 14
g/dl
  Before operation | 13.0 (1.7)
  6 months after operation | 12.5 (1.6)
  Until end of study (on average 14.8 months) | 12.5 (1.8)

9. Primary Outcome: Albumin
Description: For the evaluation of long-term safety, albumin was measured to determine malnutrition.
Time Frame: Before operation , 6 months after operation, Until end of study (on average 14.8 months)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Long Limb Roux en Y Reconstruction
Number analyzed (Participants) | 14
g/dl
  Before operation | 4.4 (0.4)
  6 months after operation | 4.3 (0.6)
  Until end of study (on average 14.8 months) | 3.9 (0.7)

10. Primary Outcome: Operation Related Mortality
Description: Operation related mortality was measured for the evaluation of safety for the operation. Operation related mortality was defined as any complication resulting in the death of the patient within 1 month or during hospitalization after operation.
Time Frame: Until end of study (on average 14.8 months)
Population: All of enrolled patient were included.(N=15)
Measure: Number; unit: participants
Groups:
- Long Limb Roux-en Y Reconstruction: Long limb Roux-en Y reconstruction means that the length of Roux limb and biliopancreatic limb are longer than conventional reconstruction method after gastrectomy.
  Until end of study (on average 14.8 months), operation related mortality of Gastric cancer patient with type 2 diabetes who receive total or Subtotal gastrectomy with long limb Roux en Y reconstruction were analyzed.
Arm/Group | Long Limb Roux-en Y Reconstruction
Number analyzed (Participants) | 15
participants | 0

11. Secondary Outcome: Matsuda Index : Good Response Group
Description: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Some patients showed normal FPG level and HbA1c < 6% without any antidiabetic medications after operation. We called this group as "good response group". We analyzed the change of insulin sensitivity after operation in good response group.
  The Matsuda index(Insulin Sensitivity Index) was obtained using the following formula:
  Matsuda index = 10000/square root of [(fasting glucose × fasting insulin) × (mean glucose × mean insulin during OGTT)]
Time Frame: Before operation , 6 months after operation, Until end of study (on average 14.8 months)
Population: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Normal FPG level and HbA1c < 6% without any antidiabetic medications were observed in 11 patients (78.6 %). We called this group as "good responder group". We analyzed the change of insulin sensitivity after operation in good responder group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Long Limb Roux-en Y Reconstruction : Good Responder Group: Long limb Roux-en Y reconstruction means that the length of Roux limb and biliopancreatic limb are longer than conventional reconstruction method after gastrectomy. Long limb Roux-en Y reconstruction : Good responder group means patients who showed normal FPG level and HbA1c < 6% without any antidiabetic medications after operation.
Arm/Group | Long Limb Roux-en Y Reconstruction : Good Responder Group
Number analyzed (Participants) | 11
units on a scale
  Before operation | 5.7 (3.0)
  6 months after operation | 14.6 (6.1)
  Until end of study (on average 14.8 months) | 12.7 (7.3)

12. Secondary Outcome: QUICKI : Good Response Group
Description: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Some patients showed normal FPG level and HbA1c < 6% without any antidiabetic medications. We called this group as "good response group". We analyzed the change of insulin sensitivity after operation in good response group. The quantitative insulin sensitivity check index (QUICKI) was measured.
  The QUICKI is obtained using the following formula:
  1 / (log(fasting insulin µU/mL) + log(fasting glucose mg/dL))
Time Frame: Before operation, 6 months after operation, Until end of study (on average 14.8 months)
Population: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Normal FPG level and HbA1c < 6% without any antidiabetic medications were observed in 11 patients (78.6 %). We called this group as "good responder group". We analyzed the change of QUICKI after operation in good responder group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Long Limb Roux-en Y Reconstruction : Good Responder Group
Number analyzed (Participants) | 11
units on a scale
  Before Operation | 0.4 (0.1)
  6 months after operation | 0.4 (0.0)
  Until end of study (on average 14.8 months) | 0.5 (0.1)

13. Secondary Outcome: HOMA-IR : Good Response Group
Description: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Some patients showed normal FPG level and HbA1c < 6% without any antidiabetic medications. We called this group as "good response group". We analyzed the change of insulin resistance after operation in good response group.
  HOMA-IR(Homeostasis model assessment-estimated insulin resistance) was measured.
  HOMA-IR was obtained using the following formula:
  Glucose(mg/dl) x Insulin/405
Time Frame: Before operation, 6 months after operation, Until end of study (on average 14.8 months)
Population: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Normal FPG level and HbA1c < 6% without any antidiabetic medications were observed in 11 patients (78.6 %). We called this group as "good responder group". We analyzed the change of HOMA-IR after operation in good responder group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Long Limb Roux-en Y Reconstruction : Good Responder Group
Number analyzed (Participants) | 11
units on a scale
  Before operation | 1.9 (1.9)
  6 months after operation | 0.9 (0.7)
  Until end of study (on average 14.8 months) | 0.8 (0.6)

14. Secondary Outcome: HOMA-B : Good Response Group
Description: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Some patients showed normal FPG level and HbA1c < 6% without any antidiabetic medications. We called this group as "good response group". We analyzed the change of beta-cell function after operation in good response group. HOMA-B(Homoeostasis model assessment-derived beta-cell function) was measured.
  HOMA-B was obtained using the following formula:
  225 × 18/fasting insulin(mU/L) × fasting glucose(mg/dL)
Time Frame: Before operation, 6 months after operation, Until end of study (on average 14.8 months)
Population: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Normal FPG level and HbA1c < 6% without any antidiabetic medications were observed in 11 patients (78.6 %). We called this group as "good responder group". We analyzed the change of beta cell function after operation in good responder group.
Measure: Mean (Standard Deviation); unit: percentage of beta cell function
Arm/Group | Long Limb Roux-en Y Reconstruction : Good Responder Group
Number analyzed (Participants) | 11
percentage of beta cell function
  Before operation | 8.7 (6.9)
  6 months after operation | 13.4 (8.9)
  Until end of study (on average 14.8 months) | 17.8 (12.3)

15. Secondary Outcome: Body Mass Index : Good Response Group
Description: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Some patients showed normal FPG level and HbA1c < 6% without any antidiabetic medications. We called this group as "good response group". We analyzed the change of weight change after operation in good response group.
  BMI(Body Mass index , kg/㎡) was measured.
  BMI was obtained using the following formula:
  Weight (kg) / (Height (m) x Height (m))
Time Frame: Before operation, 6 months after operation, Until end of study (on average 14.8 months)
Population: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Normal FPG level and HbA1c < 6% without any antidiabetic medications were observed in 11 patients (78.6 %). We called this group as "good responder group". We analyzed the change of weight after operation in good responder group.
Measure: Mean (Standard Deviation); unit: kg/㎡
Arm/Group | Long Limb Roux-en Y Reconstruction : Good Responder Group
Number analyzed (Participants) | 11
kg/㎡
  Before operation | 25.7 (3.5)
  6 months after operation | 22.0 (3.3)
  Until end of study (on average 14.8 months) | 21.5 (2.6)

16. Secondary Outcome: HbA1c : Good Response Group
Description: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Some patients showed normal FPG level and HbA1c < 6% without any antidiabetic medications. We called this group as "good response group". We analyzed the change of HbA1c after operation in good response group.
  HbA1c is formed in a non-enzymatic glycation pathway by hemoglobin's exposure to plasma glucose and measured by high-performance liquid chromatography (HPLC)
  The HbA1c was calculated as a ratio to total hemoglobin.
Time Frame: Before operation, 6 months after operation, Until end of study (on average 14.8 months)
Population: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Normal FPG level and HbA1c < 6% without any antidiabetic medications were observed in 11 patients (78.6 %). We called this group as "good responder group". We analyzed the change of HbA1c after operation in good responder group.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Long Limb Roux-en Y Reconstruction : Good Responder Group
Number analyzed (Participants) | 11
percentage of glycated hemoglobin
  Before operation | 7.2 (1.1)
  6 months after operation | 6.0 (0.5)
  Until end of study (on average 14.8 months) | 6.0 (0.6)

17. Secondary Outcome: Hemoglobin : Good Response Group
Description: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Some patients showed normal FPG level and HbA1c < 6% without any antidiabetic medications. We called this group as "good response group". For the evaluation of long-term safety, hemoglobin was measured to determine the degree of anemia and malnutrition in good response group.
Time Frame: Before operation, 6 months after operation, Until end of study (on average 14.8 months)
Population: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Normal FPG level and HbA1c < 6% without any antidiabetic medications were observed in 11 patients (78.6 %). We analyzed the change of hemoglobin after operation in good responder group for the evaluation of long-term safety.
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Long Limb Roux-en Y Reconstruction : Good Responder Group
Number analyzed (Participants) | 11
g/dl
  Before operation | 13.0 (1.7)
  6 months after operation | 12.5 (1.6)
  Until end of study (on average 14.8 months) | 12.5 (1.8)

18. Secondary Outcome: Albumin : Good Response Group
Description: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Some patients showed normal FPG level and HbA1c < 6% without any antidiabetic medications. We called this group as "good response group". We analyzed the change of albumin level after operation in good response group for the evaluation of long-term safety.
Time Frame: Before operation, 6 months after operation, Until end of study (on average 14.8 months)
Population: At the end of the study, the follow-up duration was 12.5 ± 5.5 months (6.0 - 21.7 months). Normal FPG level and HbA1c < 6% without any antidiabetic medications were observed in 11 patients (78.6 %). We analyzed the change of albumin level after operation for the evaluation of long-term safety in good responder group.
Measure: Mean (Standard Deviation); unit: g/dl
Groups:
- Long Limb Roux-en Y Reconstruction : Good Responder Group: Long limb Roux-en Y reconstruction means that the length of Roux limb and biliopancreatic limb are longer than conventional reconstruction method after gastrectomy. Long limb Roux-en Y reconstruction : Good responder group means patients who showed normal FPG level and HbA1c < 6% without any antidiabetic medications after operation.
  '
Arm/Group | Long Limb Roux-en Y Reconstruction : Good Responder Group
Number analyzed (Participants) | 11
g/dl
  Before operation | 4.4 (0.4)
  6 months after operation | 4.2 (0.6)
  Until end of study (on average 14.8 months | 3.9 (0.7)

ADVERSE EVENTS:
Time Frame: Until end of study (on average 14.8 months)
Description: Daily check up during hospitalization after operation. check up every month after discharge.
Groups:
- Long-limb Roux-en Y Reconstruction: Long limb Roux-en Y reconstruction means that the length of Roux limb and biliopancreatic limb are longer than conventional reconstruction method after gastrectomy.
Arm/Group | Long-limb Roux-en Y Reconstruction
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long-limb Roux-en Y Reconstruction (N=15)
myocardiac infart (Cardiac disorders) | 1 (1) — One had myocardial infarction treated with percutaneous transluminal coronary angioplasty with stent insertion. The patient recovered well without sequela.
dead (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — One patient had poorly differentiated neuroendocrine carcinoma, which was most aggressive gastric cancer and died due to recurrence four months after surgery. (preoperative diagnosis: poorly differentiated adenocarcinoma)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long-limb Roux-en Y Reconstruction (N=15)
Anastomosis, non-functional (morphologic abnormality) (Surgical and medical procedures) | 1 (1) — Managed with temporary stent insertion
Stricture of anastomosis of intestine (Surgical and medical procedures) | 1 (1) — Recovered with conservative management
Open wound of abdominal wall with complication (Skin and subcutaneous tissue disorders) | 1 (1) — Managed with wound closure by retension suture technique under general anesthesia.

LIMITATIONS AND CAVEATS:
One mortality due to early recurrence leading to reduced number of subject analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No